CLINICAL TRIAL: NCT03361267
Title: Comparison of Bismuth Containing Quadruple Therapy and Clarithromycin Susceptibility-based Tailored Therapy for Helicobacter Pylori First-line Eradication
Brief Title: Comparison of Bismuth Containing Quadruple Therapy and Based Tailored Therapy for H. Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Inha University Hospital, Inha University Hospital, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Inha helicobacter study
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Helicobacter Pylori Infection; Compliance, Patient; Drug Resistance; Antibiotics
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bismuth containing quadruple therapy (Active Comparator): If CLO test is positive, Bismuth containing quadruple therapy (rabeprazole 20 mg bid, metronidazole 5100 mg tid, bismuth 300 mg qid, tetracycline 500mg qid) are prescribed for 7 days If CLO test is negative, no intervention is needed
  Interventions: Diagnostic Test: CLO test
- tailored therapy (Experimental): If H. pylori PCR is negative, no intervention is needed If H. pylori PCR is positive and mutation is negative, triple regimen (rabeprazole 20 mg bid, amoxacillin 1000 mg bid, clarithromycin 500mg bid) are prescribed for 7 days is given If H. pylori PCR is positive and mutation is positive, Bismuth containing quadruple therapy (rabeprazole 20 mg bid, metronidazole 5100 mg tid, bismuth 300 mg qid, tetracycline 500mg qid) are prescribed for 7 days is given
  Interventions: Diagnostic Test: Helicobacter pylori PCR test

INTERVENTIONS:
Diagnostic Test: Helicobacter pylori PCR test — Clarithromycin resistance (-) Triple therapy (rabeprazole 20 mg bid, amoxicillin 1000mg bid, clarithromycin 500mg bid) for 7 days Clarithromycin resistance (+) Bismuth containing quadruple therapy (rabeprazole 20 mg bid, metronidazole 500 mg tid, bismuth 300 mg qid, tetracycline 500mg qid) for 7 days
  Arms: tailored therapy
Diagnostic Test: CLO test — CLO test : negative --> drop out CLO test : postive --> bismuth containing quadruple therapy
  Arms: Bismuth containing quadruple therapy

SUMMARY:
As the antibiotic resistance increases, the eradication rate of triple therapy is decreasing. Recent guideline recommend the use of bismuth-containing quadruple therapy in areas where clarithromycin resistance is greater than 15%. However, the ideal treatment would be the tailored therapy which choose the antibiotics depending on the antibiotic resistance. This study compared the eradication rates, safety and complicance of tailored therapy compared with empirical bismuth quadruple therapy in the naive patients with H. pylori infection.

DETAILED DESCRIPTION:
In order to be eligible for first-line H. pylori eradication therapy, at least 80% of eradication rate should be achieved by intention to treat (ITT) analysis. However, the triple therapy (PPI, clarithromycin, amoxicillin) is losing 1st-line therapy because of increasing antibiotic resistance. The most common cause of failure in triple therapy is clarithromycin resistance.

In the past, clarithromycin resistance was rarely observed in Korea, but the resistance rate has increased rapidly during the last 10 years, up to 37.3%.

As an alternative, Korean guidelines of Helicobacter pylori eradication in 2013 recommend that bismuth-containing antibiotics (not containing clarithromycin) should be considered in areas with high clarithromycin resistance as in Korea. However, there is a lack of research on the efficacy of bismuth-containing quadruple therapy as a 1st-line therapy. The aim of this prospectivce randomized study is to investingate the efficacy, conpliance, adverse events and cost-effectiveness between bismuth containing quadruple therapy and tailored therapy in areas with high clarithromycin resistance

ELIGIBILITY:
Inclusion Criteria:

* Participants with peptic ulcer, s/p ESD due to early gastric cancer/gastric adenoma, Maltoma
* Ability and willingness to participate in the study and to sign and give informed consent
* confirmed H. pylori infection

Exclusion Criteria:

* Previous H. pylori eradication therapy
* Less than 18 years old
* With history of H. pylori infection treatment
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs
* Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-30 (Estimated); Primary Completion 2018-06-28 (Estimated); Study Completion 2018-06-28 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test or CLO test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).
  or negative from CLO test

SECONDARY OUTCOMES:
Rate of adverse effects | within 7 days after completion of therapy
  During the 7-day treatment period, the subjects kept a diary to score any possible side effects or discomforts. The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities).
Compliance rate | within 7 days after completion of therapy
  Compliance was deﬁned as poor when they had taken less than 80% of the total medication.
Medical cost | two months after completion of therapy ]
  Summation of diagnostic fee, cost of medication and 2-line therapy cost if the 1st line therapy fails

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No